CLINICAL TRIAL: NCT03102606
Title: A Phase 3, Multicenter, Randomized, Double Blind, Study to Evaluate Duration of Severe Neutropenia With Plinabulin Versus Pegfilgrastim in Patients With Solid Tumors Receiving Docetaxel Myelosuppressive Chemotherapy (Protective 1)
Brief Title: Plinabulin vs. Pegfilgrastim in Patients With Solid Tumors Receiving Docetaxel Myelosuppressive Chemotherapy Phase 3
Acronym: Protective-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeyondSpring Pharmaceuticals Inc. (Industry)
Collaborators: Covance (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BPI-2358-105 phase 3
Record Dates: First submitted 2017-03-06; First posted 2017-04-06 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Neutropenia
Keywords: Plinabulin; Pegfilgrastim; Duration of Severe Neutropenia; Bone Pain
MeSH Terms: interventions — NPI 2358; pegfilgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Plinabulin and pegfilgrastim are each masked using a double-dummy design in phase 3.
  Docetaxel administration is not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel (75 mg/m2) + pegfilgrastim (6 mg) + placebo matching plinabulin (Active Comparator): Arm 1
  Interventions: Drug: Pegfilgrastim; Other: D5W Placebo
- Docetaxel (75 mg/m2) + plinabulin (40 mg) + placebo matching pegfilgrastim (Experimental): Arm 2
  Interventions: Drug: Plinabulin; Other: Saline Placebo

INTERVENTIONS:
Drug: Plinabulin — Plinabulin (BPI-2358) is a synthetic, low molecular weight, new chemical entity that belongs to the diketopiperazine class of compounds. Plinabulin is intended for intravenous (IV) infusion and is diluted in D5W and administered for 30 minutes (± 5 minutes).
  Other Names: BPI-2358; NPI-2358
  Arms: Docetaxel (75 mg/m2) + plinabulin (40 mg) + placebo matching pegfilgrastim
Drug: Pegfilgrastim — PEGFILGRASTIM is a long-acting granulocyte colony-stimulating factor that stimulates the growth of neutrophils, to reduce the incidence of fever and infection in patients with certain types of cancer who are receiving chemotherapy that affects the bone marrow.
  Other Names: Neulasta; G-CSF
  Arms: Docetaxel (75 mg/m2) + pegfilgrastim (6 mg) + placebo matching plinabulin
Other: Saline Placebo — Placebo Syringe 0.6 ml Saline to match the 0.6 ml pegfilgrastim administration
  Arms: Docetaxel (75 mg/m2) + plinabulin (40 mg) + placebo matching pegfilgrastim
Other: D5W Placebo — Placebo 250 ml D5W to match the administration of plinabulin diluted in 250 ml D5W
  Arms: Docetaxel (75 mg/m2) + pegfilgrastim (6 mg) + placebo matching plinabulin

SUMMARY:
To assess Duration of Severe Neutropenia (DSN) in treatment Cycle 1 in patients with advanced or metastatic breast cancer, who have failed >/= 1 but < 5 prior lines of chemotherapy; locally advanced or metastatic non small cell lung cancer (NSCLC) after platinum therapy failure; or hormone refractory (androgen independent) metastatic prostate cancer treated with docetaxel (75 mg/m2) + plinabulin (40 mg) versus docetaxel (75 mg/m2) + pegfilgrastim (6 mg). Neutrophils count will be assessed at baseline; Pre dose during Cycle 1, Day 1, 2, 6, 7, 8, 9, 10, 15.

*Study is officially closed on 08 Feb 2021*

DETAILED DESCRIPTION:
Arm 1: Docetaxel (75 mg/m2) + pegfilgrastim (6 mg) + placebo matching plinabulin

Arm 2: Docetaxel (75 mg/m2) + plinabulin (40 mg) + placebo matching pegfilgrastim

ELIGIBILITY:
Inclusion Criteria:

1. At least ≥ 18 years of age (male or female) at the time of signing the informed consent form.
2. ECOG performance status of 0 to 1.
3. Patients with:

   Phase 2 only:

   • Advanced or metastatic NSCLC failing platinum-based therapy

   Phase 3 only:
   * Advanced or metastatic breast cancer, who have failed < 5 prior lines of chemotherapy (Note that study treatment may be the first chemotherapy treatment for advanced or metastatic cancer)
   * locally advanced or metastatic NSCLC after platinum therapy failure
   * HRPC (Note that study treatment may be the first chemotherapy treatment)
4. Pathology confirmation of cancer is required.
5. Patients with ≥ 1 of the following risk factors, at the initiation of docetaxel chemotherapy, that would require neutropenia prophylaxis per National Comprehensive Cancer Network (NCCN) guidelines (version 2, 2016):

   * Prior chemotherapy or radiation treatment
   * Bone marrow involvement by tumor
   * Surgery and/or open wounds within 4 weeks of first administration of study drug
   * Age > 65 years of age and receiving full chemotherapy dose intensity
6. Life expectancy of 3 months or more.
7. The following laboratory results assessed within 14 days prior to study drug administration:

   * Hemoglobin >/= 9 g/dL independent of transfusion or growth factor support
   * Absolute neutrophil count (ANC) >/= 1.5 x 10**9/L independent of growth factor support
   * Serum total bilirubin </= 1.5 times the upper limit normal (ULN), unless the patient has a diagnosis of Gilbert's disease, in which case direct bilirubin </= 1.5 times ULN of the direct bilirubin.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) </= 2.5 x ULN (</= 1.5 x ULN if alkaline phosphatase is > 2.5 x ULN)
   * Serum creatinine </= 1.5 x ULN

   Note: Results are from the central laboratory. Local laboratory results may be accepted on a case by case basis after discussion with the Medical Monitor, however in this case central laboratories must also be taken within the screening time window.
8. Prothrombin time (PT)/International Normalized Ratio (INR) ≤ 1.5 × upper limit of normal (ULN), activated partial thromboplastin time (PTT) ≤ 1.5 × ULN, based on central laboratory results.
9. Female subjects of childbearing potential have a negative pregnancy test at screening. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

   * Women of childbearing potential (i.e., menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.
   * Sexually active women of childbearing potential enrolled in the study must agree to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner.
   * For male patients who are sexually active and who are partners of premenopausal women: agreement to use two forms of contraception during the treatment period and for at least 3 months after the last dose of study drug.

Exclusion Criteria:

1. History of myelogenous leukemia, myelodysplastic syndrome or concomitant sickle cell disease.
2. Received chemotherapy within 4 weeks prior to the first dose of study drug.
3. Received prior docetaxel treatment, except adjuvant docetaxel given > 1 year prior to first dose of study drug
4. Phase 3 only: Received >/= 5 lines of cytotoxic chemotherapy for advanced or metastatic breast cancer (adjuvant chemotherapy will count as one line of chemotherapy, and any hormonal or biological, non conjugate therapy [e.g., trastuzumab] will not count as a line of therapy).
5. Current use of strong cytochrome P450 (CYP) 3A4 inhibitors, within 3 days of the first administration of study drug, and 7 days after treatment with taxanes OR requires use of strong CYP3A4 inhibitors
6. Received an investigational agent or tumor vaccine within 2 weeks before the first dose of study drug; patients must have recovered from toxicity of prior treatment and have no > Grade 1 CTCAE (v4.03) treatment emergent AEs.
7. Receiving any concurrent anticancer therapies (except continued hormonal treatment).
8. Received a prior bone marrow or stem cell transplant.
9. Has a co-existing active infection or received systemic anti-infective treatment within 72 hours before the first dose of study drug.
10. Prior radiation therapy within the 4 weeks before the first dose of study drug.
11. Prior use of pegfilgrastim or filgrastim within 4 weeks before the first dose of study drug.
12. Presence of any serious or uncontrolled illness including, but not limited to: uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled arterial thrombosis, symptomatic pulmonary embolism, or psychiatric illness that would limit compliance with study requirements, or any other conditions that would preclude the patient from study treatment as per the discretion of the Investigator.
13. Significant cardiovascular history:

    * History of myocardial infarction or ischemic heart disease within 1 year (within a window of up to 18 days less than 1 year) before first study drug administration;
    * Uncontrolled arrhythmia;
    * History of congenital QT prolongation;
    * Electrocardiogram (ECG) findings consistent with active ischemic heart disease;
    * New York Heart Association Class III or IV cardiac disease;
    * Uncontrolled hypertension: blood pressure consistently >150 mm Hg systolic and > 100 mm Hg diastolic in spite of antihypertensive medication.
14. History of hemorrhagic diarrhea, inflammatory bowel disease, or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
15. Any other malignancy requiring active therapy.
16. Known human immunodeficiency virus (HIV) seropositivity.
17. Active Hepatitis B virus (HBV) infection which requires antiviral treatment. Patients with detectable Hepatitis B surface Antigen (HBsAg) may be eligible provided the patient has a negative viral load. Patients with a positive HBsAg must have a negative viral load before each chemotherapy administration. Hepatitis B surface antibody (anti HBs) without detectable HBsAg does NOT exclude patients from the study. Hepatitis C infection (Hepatitis C antibody reactive) which requires treatment also excludes patients from the study.
18. Female subject who is pregnant or lactating.
19. Unwilling or unable to comply with procedures required in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Blayney, MD, Principal Investigator — Stanford University School of Medicine - Cancer Institute
Locations (18):
- United States (3):
  - Stanford University School of Medicine - Cancer Institute, Stanford, California
  - Hematology/Oncology of the North Shore, Skokie, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
- China (6):
  - Heilongjiang Cancer Hospital, Harbin, Heilongjiang
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Linyi Cancer Hospital, Linyi
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Henan Cancer Hospital, Zhengzhou
- Russia (3):
  - State Budgetary Healthcare Institution of Stavropol Territory "Pyatigorsk Interregional Oncology Dispensary", Pyatigorsk
  - SBI of Healthcare "Oncology Dispensary #2" Ministry of Healthcare of Krasnodar Region, Sochi
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
- Ukraine (6):
  - Dnipropetrovsk City Multifunctional Hospital, Dnipro
  - Prykarpatskiy Regional Oncological Center, Ivano-Frankivsk
  - Communal Institution of Kherson Regional Council "Kherson regional oncological dispensary", Kherson
  - Kryvyi Rih Oncology Dispensary, Kryvyi Rih
  - Lviv State Oncological Regional Treatment and Preventive Center, Lviv
  - Municipal Institution "Sumy Regional Clinical Oncology Dispensary", Sumy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blayney DW, Mohanlal R, Adamchuk H, Kirtbaya DV, Chen M, Du L, Ogenstad S, Ginn G, Huang L, Zhang Q. Efficacy of Plinabulin vs Pegfilgrastim for Prevention of Docetaxel-Induced Neutropenia in Patients With Solid Tumors: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2145446. doi: 10.1001/jamanetworkopen.2021.45446. PMID 35084480
- [Derived] Blayney DW, Zhang Q, Feng J, Zhao Y, Bondarenko I, Vynnychenko I, Kovalenko N, Nair S, Ibrahim E, Udovista DP, Mohanlal R, Ogenstad S, Ette E, Du L, Huang L, Shi YK. Efficacy of Plinabulin vs Pegfilgrastim for Prevention of Chemotherapy-Induced Neutropenia in Adults With Non-Small Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):e204429. doi: 10.1001/jamaoncol.2020.4429. Epub 2020 Nov 12. PMID 32970104

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Started | 53 | 52
Completed | 39 | 45
Not Completed | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 40 | 74
  >=65 years | 19 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.85) | 57.0 (10.79) | 58.0 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 21 | 19 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 25 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Neutropenia (DSN)
Description: Duration of severe neutropenia (ANC < 0.5 × 109/L)
Time Frame: 21 Days
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Days | 0.246 [0.205 to 0.287] | 0.770 [0.682 to 0.857]

2. Secondary Outcome: Change in Estimated Mean Bone Pain Score
Description: Change in estimated mean bone pain score from pre-dose Day 1 through Day 8. The bone pain scale assessment was based on the validated Wong-Baker Faces® Pain Rating Scale. The pain scale range is from 0 to 10. The severity of pain marked on a scale is from 0 ('no hurt') to 10 ('hurt worst').
Time Frame: Day 1 through 8 in Cycle 1 (each cycle is 21 days)
Measure: Least Squares Mean (Standard Error); unit: Wong-Baker FACES Pain Scale (range:0-10)
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Wong-Baker FACES Pain Scale (range:0-10) | 2.35 (0.178) | 1.69 (0.179)

3. Secondary Outcome: Change in Patients With at Least 30% Platelet Count From Baseline in Cycle 1
Description: Patients with platelet count at least 30% change from baseline at any time during Cycle 1
Time Frame: Anytime during Cycle 1 (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Participants | 41 | 23

4. Secondary Outcome: Proportion of Patients With Neutrophil-to-lymphocyte Ratio (NLR) > 5
Description: Proportion of patients with neutrophil-to-lymphocyte ratio (NLR) > 5 from Day 1 through Day 15
Time Frame: 15 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Participants | 24 | 2

5. Secondary Outcome: Proportion of Patients With Thrombocytopenia
Description: Proportion of patients with thrombocytopenia (all grade) during 4 cycles
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Participants | 19 | 10

6. Secondary Outcome: Infections
Description: Incidence of infections in cycles 1 to 4
Time Frame: 84 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Participants | 8 | 4

7. Secondary Outcome: Antibiotic Use
Description: Incidence of antibiotic use
Time Frame: 21 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Participants | 7 | 8

8. Secondary Outcome: Sepsis
Description: To assess the incidence of sepsis
Time Frame: 84 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
Number analyzed (Participants) | 53 | 52
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim
All-Cause Mortality (participants affected / at risk) | 1/53 | 2/52
Serious Adverse Events (participants affected / at risk) | 6/53 | 8/52
Other Adverse Events (participants affected / at risk) | 49/53 | 51/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin (N=53) | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim (N=52)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 2/2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel (75 mg/m2) + Pegfilgrastim (6 mg) + Placebo Matching Plinabulin (N=53) | Docetaxel (75 mg/m2) + Plinabulin (40 mg) + Placebo Matching Pegfilgrastim (N=52)
Anemia (Blood and lymphatic system disorders) | 13 | 17
Neutropenia (Blood and lymphatic system disorders) | 7 | 12
Leukopenia (Blood and lymphatic system disorders) | 7 | 10
Tachycardia (Cardiac disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 11
Nausea (Gastrointestinal disorders) | 8 | 8
Constipation (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 10 | 7
Malaise (General disorders) | 5 | 9
Fatigue (General disorders) | 2 | 6
Pyrexia (General disorders) | 2 | 3
Face oedema (Gastrointestinal disorders) | 1 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 4
Neutrophil count decreased (Investigations) | 10 | 23
White blood cell count decreased (Investigations) | 10 | 21
Alanine aminotransferase increased (Injury, poisoning and procedural complications) | 8 | 7
Aspartate aminotransferase increased (Investigations) | 8 | 7
Platelet count decreased (Investigations) | 6 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 8
Decreased appetite (Metabolism and nutrition disorders) | 5 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 17
Hypertension (Vascular disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT03102606/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT03102606/SAP_001.pdf